CLINICAL TRIAL: NCT01745965
Title: A Prospective, Randomized Multicenter, Open-label Comparison of Preoperative Trastuzumab Emtansine (T-DM1) With or Without Standard Endocrine Therapy vs. Trastuzumab With Standard Endocrine Therapy Given for Twelve Weeks in Patients With Operable HER2+/HR+ Breast Cancer Within the ADAPT Protocol.
Acronym: ADAPT; T-DM1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM06/ADAPT HER2+/HR+
Record Dates: First submitted 2012-11-30; First posted 2012-12-10 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T-DM1 (Experimental): single agent T-DM1 for 12 weeks (3,6 mg/kg q3w)
  Interventions: Drug: T-DM1
- T-DM1 + endocrine therapy (Experimental): Single agent T-DM1 for 12 weeks (3,6 mg/kg q3w) with standard endocrine therapy (tamoxifen in premenopausal women and an aromatase inhibitor in postmenopausal women, if no contraindications are present, in a standard daily dosage).
  Interventions: Drug: T-DM1
- Trastuzumab + endocrine therapy (Active Comparator): The control group will receive trastuzumab in 3-weekly schedule (8 mg/kg as loading dose and then 6 mg/kg q3w)with endocrine therapy tamoxifen in premenopausal women and an aromatase inhibitor in postmenopausal women, if not contraindications are present, in a standard daily dosage).
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: T-DM1
  Arms: T-DM1; T-DM1 + endocrine therapy
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Trastuzumab + endocrine therapy

SUMMARY:
Trial to optimize neoadjuvant therapy for HER overexpression and co-expressing of hormone receptors(ER and/or PR) breast cancer (HEr2+/HR+).

A new high potential trastuzumab conjugate T-DM1(trastuzumab was linked with the cytotoxic agent mertansine DM1)was tested with endocrine therapy and without against a standard arm with trastuzumab and endocrine therapy.

DETAILED DESCRIPTION:
the neoadjuvant therapy Patients with HER2+/HR+ (HER2+ and ER+ and/or PR+) tumor will receive single agent T-DM1 for 12 weeks (3,6 mg/kg q3w) with or without standard endocrine therapy (tamoxifen in premenopausal women and an aromatase inhibitor in postmenopausal women, if not contraindications are present, in a standard daily dosage). The control group will receive trastuzumab in 3-weekly schedule (8 mg/kg as loading dose and then 6 mg/kg q3w) in combination with the same standard endocrine therapy, if no contraindications are existent.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 years and above (consider patients at 70 years and above for ADAPT Elderly)
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1 - T4 (except inflammatory breast cancer)
* All clinical N (cN)
* No clinical evidence for distant metastasis (M0)
* Known HR status and HER2 status (local pathology) Tumor block available for central pathology review
* Performance Status ECOG ≤ 1 or KI ≥ 80%
* Negative pregnancy test (urine or serum) within 7 days prior to start of induction treatment in premenopausal patients
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up

Additional Inclusion criteria for participation in the HER2+/HR+ sub-protocol:

* Confirmed ER and/or PR positive and HER2+ by central pathology
* Clinical cT1c - T4a-c (participation of patients with tumors >cT2 is strongly recommended)
* All clinical N (participation of patients with cN0, if cT1c is strongly recommended)
* Patients must qualify for neoadjuvant treatment
* LVEF > 50%; LVEF within normal limits of each institution measured by echocardiography and normal ECG (within 42 days prior to induction treatment)

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin, pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry
* Male breast cancer
* Concurrent pregnancy; patients of childbearing potential must implement
* a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Reasons indicating risk of poor compliance Patient not able to consent

Additional Exclusion Criteria for participation in the HER2+/HR+ sub-protocol:

* Known polyneuropathy ≥ grade 2
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study
* Inadequate organ function (e.g. hepatic impairment, pulmonary disease, etc.)
* Uncompensated cardiac function (current unstable ventricular arrhythmia
* requiring treatment, history of symptomatic CHF NYHA classes II-IV), history of myocardial infarction or unstable angina pectoris within 6 months of enrollment, history of severe hypertension, CAD - coronary artery disease)
* Severe dyspnea
* Pneumonitis

Abnormal blood values:

* Thrombocytopenia > CTCAE grade 1
* Increases in ALT/AST > CTCAE grade 1
* Hypokalaemia > CTCAE grade 1
* Neutropenia > CTCAE grade 1
* Anaemia > CTCAE grade 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the pCR rates in patients with HER2+/HR+ breast cancer treated by preoperative T-DM1 with or without standard endocrine therapy or trastuzumab with endocrine therapy. | After 12 weeks
  pCR will be measured after 12 weeks of randomized treatment.
Evaluation of dynamic testing (based on proliferation/apoptosis changes in serial biopsy and imaging by MRI) after three weeks of treatment as a surrogate parameter for response. | after 3 weeks of treamtment
  Response: pCR (residual cancer burden (RCB) 0-1) or resistance/low response (RCB II-III or progressive disease)

SECONDARY OUTCOMES:
Evaluation of dynamic test regarding prediction of 5-year event-free survival (EFS) | 5 year after treatment
Overall survival | 5 year after treamtment
Toxicity/cardiac safety | 5 years after treatment
Overall safety in the three treatment arms | 5 years after treatment
Health-related quality of life (HRQL) | After 5 year after treatment of last patient

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Center of the University of Munich (LMU), Universitätsfrauenklinik Großhadern, Munich, Germany; Ulrike Nitz, Prof. Dr., Study Chair — Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany
Locations (2):
- Germany (2):
  - Ev. Krankenhaus Bethesda Brustzentrum Niederrhien, Mönchengladbach
  - Breast Center of the University of Munich (LMU), Munich

REFERENCES:
- [Background] Hofmann D, Nitz U, Gluz O, Kates RE, Schinkoethe T, Staib P, Harbeck N. WSG ADAPT - adjuvant dynamic marker-adjusted personalized therapy trial optimizing risk assessment and therapy response prediction in early breast cancer: study protocol for a prospective, multi-center, controlled, non-blinded, randomized, investigator initiated phase II/III trial. Trials. 2013 Aug 19;14:261. doi: 10.1186/1745-6215-14-261. PMID 23958221